CLINICAL TRIAL: NCT06508528
Title: A 12-week Growth Mindset Intervention for Intern Nursing Students
Brief Title: Intervention of Growth Mindset for Intern Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huzhou University (Other)
Collaborators: Hangzhou Normal University (Other); The Affiliated Hospital of Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Hailu Wu, master, Huzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022032
Record Dates: First submitted 2024-07-13; First posted 2024-07-18 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Growth, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth mindset intervention group (Experimental): Internship nursing students received a 12-week growth mindset intervention.
  Interventions: Behavioral: a 12-week growth mindset intervention
- Hospital Teaching Team (Other): Controlled group will receive regular hospital teaching.
  Interventions: Other: Hospital mentoring

INTERVENTIONS:
Behavioral: a 12-week growth mindset intervention — This is a 12-week growth mindset intervention for the nursing students during clinical rotation practice. It aims at promoting the core self-evaluation and professional sefl-efficacy for them. The intervention has 12 themes, with each intervention lasting 15 to 20 minutes. Intervention will be carried out through a combination of online and offline methods.
  Arms: Growth mindset intervention group
Other: Hospital mentoring — The control group will receive guidance from the hospital. Including self-regulation of stress, self-protection in clinical practice, and so on
  Arms: Hospital Teaching Team

SUMMARY:
This is a 12-week growth mindset intervention for the nursing students during clinical rotation practice. It aims at promoting the core self-evaluation and professional self-efficacy for them.

DETAILED DESCRIPTION:
64 intern nursing students from a hospital in China were recruited for this study and randomly assigned to the intervention group and control group.

ELIGIBILITY:
Inclusion Criteria:

* full-time intern nursing students including Junior college and undergraduate students；
* require a clinical nursing internship for at least 8 months ；
* know the purpose of the study and volunteer to participate in the study.

Exclusion Criteria:

* recently experienced significant stress events such as accidental injuries, nursing accidents, etc；
* receiving other training that may affect this intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

PRIMARY OUTCOMES:
growth mindset | We will measure the score of growth mindset before the training, 6 weeks of training, and 12 weeks of training.
  Growth mindset in recent one week measured by the growth mindset scale , ranging from 6-36, with higher score reflects higher level of growth mindset.
core self-evaluation | We will measure the score of core self-evaluation before the training, 6 weeks of training, and 12 weeks of training.
  Core self-evaluation in recent one week measured by the core self-evaluation scale, ranging from 10-50, with higher score reflects higher level of core self-evaluation.
professional self-efficacy | We will measure the score of professional self-efficacy before the training, 6 weeks of training, and 12 weeks of training.
  Professional self-efficacy in recent one week measured by the professional self-efficacy questionnaire for nursing students, ranging from 27-135, with higher score reflects higher level of professional self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: MeiJuan Cao, Dr., Study Director — Huzhou University
Locations (1):
- Hangzhou Normal University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No
The participants are not willing to share the data.